CLINICAL TRIAL: NCT06385431
Title: Obeservational Cohort for Evaluating Future Cardiovascular Disease With High Metabolic Risks
Acronym: Charm
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiangqing Kong, director of the department of cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: Charm
Record Dates: First submitted 2024-04-09; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cardiovascular and metabolic disease
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — obeservational study with none intervention

SUMMARY:
Cardiovascular and metabolic diseases refer to a large category of cardiovascular diseases accompanied by a series of metabolic disorders (including dyslipidemia, obesity, abnormal glucose tolerance, diabetes, hypertension, thyroid dysfunction, etc.), which is the primary cause of death and disease burden of Chinese residents.The number of deaths from atherosclerotic cardiovascular disease (ASCVD) in China is about 2.4 million, accounting for 61% of the total cardiovascular deaths, accounting for more than 40% of the all-cause deaths. In Chinese patients with coronary heart disease, 52.9% are complicated with diabetes.Despite the 1.1 million coronary stents implanted in China, there has been no reduction in cardiovascular mortality, which highlights the importance of threshold advancement and the management of metabolic risk factors.

In recent years, the new concept of cardiovascular and metabolic diseases has been actively promoted at home and abroad, and the focus of prevention and treatment strategy of cardiovascular and metabolic diseases has been called for.The project proposed the concept of co-treatment of metabolic diseases based on disorders of blood pressure regulation, disorders of glucose metabolism and disorders of lipid metabolism. Subjects eligible for cardiovascular and metabolic diseases were screened, their past medical records were registered, education and diagnosis and treatment management were conducted.

ELIGIBILITY:
Inclusion Criteria:

1.18 years old ≤ age ≤70 years old; 2. Have ≥1 cardiovascular and metabolic disease:

1. hypertension (systolic blood pressure ≥140mmHg in the resting room and diastolic blood pressure ≥90mmHg in the rest room;Previously diagnosed and taking blood pressure medication);
2. Dyslipidemia: [LDL-C≥4.1mmol/L and/or HDL-C<1.0mmol/L and/or TC≥6.2mmol/L and/or TG≥2.3mmol/L];
3. fatty liver;
4. Obesity (BMI≥28kg/m2 or waist circumference: male ≥90cm, female ≥85cm);
5. Abnormal glucose metabolism:

Impaired fasting blood glucose: fasting blood glucose ≥6.1, <7.0mmol/L, 2h post-glucose load blood glucose<7.8mmol/L And/or impaired glucose tolerance: fasting blood glucose<6.1mmol/L, 2h post-glucose load blood glucose ≥7.8,<11.1mmol/L and/or HbA1c≥5.7, <6.5%; 3. Subjects voluntarily participate in the study

Exclusion Criteria:

1. Diagnosed type 1 and/or type 2 diabetes;
2. Confirmed history of secondary hypertension (renal parenchymatous hypertension, renal artery stenosis, primary aldosteronism, pheochromocytoma, Cushing's syndrome, coarctation of the aorta, obstructive sleep apnea hypopnea syndrome, etc.);
3. A history of malignant tumors (other than non-metastatic skin basal cell carcinoma or squamous cell carcinoma or cervical cancer in situ that has been appropriately treated or resected);
4. Severe structural heart disease (including valvular heart disease, cardiomyopathy, congenital heart disease);
5. Myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack in the last 6 months;
6. History of cardiovascular and cerebrovascular surgery/interventional treatment (stent, balloon, thrombectomy, etc.);
7. Pregnant women or those who are breastfeeding;
8. Patients with clear immune system abnormalities (systemic lupus erythematosus, etc.);
9. Impaired liver and kidney function (ALT, AST more than 3 times the upper limit of normal, eGFR(CKD-EPI)≤60 mL/min/1.73m2);
10. Patients who cannot follow through on screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants were patients aged 18-70 years with cardiovascular and metabolic disease
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-04-28 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
incidence rate of cardiovascular and metabolic diseases | 2024.04-2026.04
  Describe the incidence rate of cardiovascular and metabolic diseases(%).
treatment rate of cardiovascular and metabolic diseases | 2024.04-2026.04
  Describe the treatment rate of cardiovascular and metabolic diseases(%)：the number of subjects with treatment/number of all subjects
control rate of cardiovascular and metabolic diseases. | 2024.04-2026.04
  Describe the control rate of cardiovascular and metabolic diseases. (%) number of subjects with effective treatment/ number of subjects with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqing Kong, Phd, Study Director — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No